CLINICAL TRIAL: NCT00309634
Title: Observer-blind Monocentric Study in Adults Aged Between 18-60 Years to Evaluate Reactogenicity and Immunogenicity of 1 and 2 Administrations of Pandemic Monovalent Influenza Vaccines Administered at Different Antigen Doses and Adjuvanted or Not
Brief Title: Study to Evaluate the Safety and Immunogenicity of a Pandemic Influenza Vaccine in Adults Aged Between 18 and 60 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: 106750
Record Dates: First submitted 2006-03-31; First posted 2006-04-03 (Estimated); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: prophylaxis of pandemic influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: 4 adjuvanted pandemic influenza candidate vaccines
Biological: 4 non-adjuvanted pandemic influenza candidate vaccines
  Other Names: 4 adjuvanted pandemic influenza candidate vaccines

SUMMARY:
Today, the leading contender for the next pandemic of influenza is H5N1, a strain of avian virus. Prevention and control of a pandemic will depend on the rapid production and worldwide distribution of specific pandemic vaccines. Candidate 'pandemic-like' vaccines must be developed and tested in clinical trials to determine the most optimal formulation and the best vaccination schedule.This study is designed to test in healthy adults aged between 18-60 years the reactogenicity and immunogenicity of one and two administrations of a candidate pandemic H5N1 vaccine formulated from Split Virus. The vaccines contain different antigen doses . For each dose, adjuvanted vaccine will be compared to the plain vaccine in order to detect the optimal formulation for immunization against the H5N1 influenza strain.

ELIGIBILITY:
Inclusion criteria:

* A male or female between, and including, 18 and 60 years of age at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential.

Exclusion criteria:

* Administration of any vaccine during the period starting 15 days before the first administration of the study vaccine and ending 21 after the second one.
* Administration of an influenza vaccine other than the study vaccines during the entire study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first administration of the study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination
* History of hypersensitivity to vaccines.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Acute clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first administration of the study vaccine or during the study.
* lactating women
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days prior to the first vaccination, or planned use during the study period.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2006-03-27 (Actual); Primary Completion 2006-10-28 (Actual); Study Completion 2006-10-28 (Actual)

PRIMARY OUTCOMES:
To evaluate the humoral immune response induced by the study vaccines in term of anti-haemagglutinin antibody titers.
To evaluate the safety and reactogenicity of the study vaccines in term of solicited local and general adverse events, unsolicited adverse events and serious adverse events"

SECONDARY OUTCOMES:
To evaluate the humoral immune response induced by the study vaccines in term of serum neutralizing antibody titers
To evaluate the cell-mediated immune response induced by the study vaccines in term of frequency of influenza-specific CD4/CD8 T lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Leroux-Roels I, Bernhard R, Gerard P, Drame M, Hanon E, Leroux-Roels G. Broad Clade 2 cross-reactive immunity induced by an adjuvanted clade 1 rH5N1 pandemic influenza vaccine. PLoS One. 2008 Feb 27;3(2):e1665. doi: 10.1371/journal.pone.0001665. PMID 18301743
- [Derived] Leroux-Roels I, Borkowski A, Vanwolleghem T, Drame M, Clement F, Hons E, Devaster JM, Leroux-Roels G. Antigen sparing and cross-reactive immunity with an adjuvanted rH5N1 prototype pandemic influenza vaccine: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):580-9. doi: 10.1016/S0140-6736(07)61297-5. PMID 17707753
- See also: Results for study 106750 can be found on the GSK Clinical Study Register — https://www.gsk-clinicalstudyregister.com/study/106750?search=study&b%22b''%22#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 106750 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106750 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 106750 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 106750 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 106750 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 106750 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register